CLINICAL TRIAL: NCT04436523
Title: Outcomes of Blood Flow Restriction Training in Post-operative Rehabilitation After Meniscus Repair Surgery
Brief Title: Blood Flow Restriction After Meniscus Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-29641
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Meniscus Disorder; Meniscus, Torn Tibial; Meniscus Lesion; Meniscus Tear, Tibial; Atrophy, Muscular
Keywords: blood flow restriction; rehabilitation; meniscus repair
MeSH Terms: conditions — Tibial Meniscus Injuries; Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Blood flow restriction (Experimental): The blood flow restriction arm will include the use of the pneumatic tourniquet applied to the operative lower extremity throughout post-operative rehabilitation sessions. The tourniquet pressure will be titrated to 80% of the measured extremity arterial limb occlusion pressure with the participant lying supine.
  Interventions: Device: Blood flow restriction (Delfi Personalized Tourniquet System); Other: Standard rehabilitation
- Standard rehabilitation (Sham Comparator): The standard rehabilitation arm will undergo the same rehabilitation protocol as the experimental arm. A tourniquet will still be applied, but will only be inflated to 20 mmHg, a pressure that will not occlude blood flow.
  Interventions: Other: Standard rehabilitation

INTERVENTIONS:
Device: Blood flow restriction (Delfi Personalized Tourniquet System) — The Delfi Personalized Tourniquet System will be utilized to apply the blood flow restriction protocol.
  Other Names: Delfi Personalized Tourniquet System
  Arms: Blood flow restriction
Other: Standard rehabilitation — Post-operative physical therapy as guided by a standardized protocol for patients undergoing meniscus repair.

SUMMARY:
The purpose of this study is to evaluate post-operative outcomes after meniscus surgery in participants undergoing blood flow restriction training as a rehabilitative adjunct compared to those with standard rehabilitation.

DETAILED DESCRIPTION:
The investigators will conduct a double-blinded, single-institution, randomized controlled trial to compare patients undergoing arthroscopic meniscus repair with post-operative rehabilitation protocol as (1) a standard-of-care rehabilitative protocol with a non-occlusive blood pressure cuff (inflated to 20-30 mm Hg) applied to the operative extremity versus (2) blood flow restriction training with cuff occlusion applied to the operative extremity. Patients will be enrolled prospectively and pre-operatively at their initial clinic visit after meniscus injury.

Rehabilitative exercises would be advanced per the physical therapists' discretion with similar exercises for patients in both groups for direct comparison. These exercises are part of an already-established post-operative protocol that is in place, with the only difference being the addition of the blood flow restriction protocol in the intervention group. All patients would undergo their supervised post-operative rehabilitation at our institution.

ELIGIBILITY:
Inclusion Criteria:

* Participants who undergo surgery for arthroscopic meniscus repair

Exclusion Criteria:

* Participants undergoing surgery for concomitant ligamentous surgeries
* Patients with Diabetes Mellitus, vascular disease, or infections of the involved extremity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee extension torque at Week 1 | Week 1 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Peak knee extension torque (Newton-meters/kilogram) evaluated with a hand-held dynamometer
Knee extension torque at Week 2 | Week 2 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Peak knee extension torque (Newton-meters/kilogram) evaluated with a hand-held dynamometer
Knee extension torque at Week 3 | Week 3 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Peak knee extension torque (Newton-meters/kilogram) evaluated with a hand-held dynamometer
Knee extension torque at Week 4 | Week 4 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Peak knee extension torque (Newton-meters/kilogram) evaluated with a hand-held dynamometer
Knee extension torque at Week 5 | Week 5 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Peak knee extension torque (Newton-meters/kilogram) evaluated with a hand-held dynamometer
Knee extension torque at Week 6 | Week 6 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Peak knee extension torque (Newton-meters/kilogram) evaluated with a hand-held dynamometer
Knee extension torque at Week 7 | Week 7 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Peak knee extension torque (Newton-meters/kilogram) evaluated with a hand-held dynamometer
Knee extension torque at Week 8 | Week 8 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Peak knee extension torque (Newton-meters/kilogram) evaluated with a hand-held dynamometer
Knee extension torque at Week 9 | Week 9 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Peak knee extension torque (Newton-meters/kilogram) evaluated with a hand-held dynamometer
Knee extension torque at Week 10 | Week 10 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Peak knee extension torque (Newton-meters/kilogram) evaluated with a hand-held dynamometer
Knee extension torque at Week 11 | Week 11 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Peak knee extension torque (Newton-meters/kilogram) evaluated with a hand-held dynamometer
Knee extension torque at Week 12 | Week 12 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Peak knee extension torque (Newton-meters/kilogram) evaluated with a hand-held dynamometer
Thigh circumference at Week 1 | Week 1 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Measurement of thigh circumference (centimeters) will be performed utilizing tape measures at specified distances along the thigh
Thigh circumference at Week 2 | Week 2 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Measurement of thigh circumference (centimeters) will be performed utilizing tape measures at specified distances along the thigh
Thigh circumference at Week 3 | Week 3 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Measurement of thigh circumference (centimeters) will be performed utilizing tape measures at specified distances along the thigh
Thigh circumference at Week 4 | Week 4 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Measurement of thigh circumference (centimeters) will be performed utilizing tape measures at specified distances along the thigh
Thigh circumference at Week 5 | Week 5 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Measurement of thigh circumference (centimeters) will be performed utilizing tape measures at specified distances along the thigh
Thigh circumference at Week 6 | Week 6 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Measurement of thigh circumference (centimeters) will be performed utilizing tape measures at specified distances along the thigh
Thigh circumference at Week 7 | Week 7 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Measurement of thigh circumference (centimeters) will be performed utilizing tape measures at specified distances along the thigh
Thigh circumference at Week 8 | Week 8 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Measurement of thigh circumference (centimeters) will be performed utilizing tape measures at specified distances along the thigh
Thigh circumference at Week 9 | Week 9 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Measurement of thigh circumference (centimeters) will be performed utilizing tape measures at specified distances along the thigh
Thigh circumference at Week 10 | Week 10 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Measurement of thigh circumference (centimeters) will be performed utilizing tape measures at specified distances along the thigh
Thigh circumference at Week 11 | Week 11 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Measurement of thigh circumference (centimeters) will be performed utilizing tape measures at specified distances along the thigh
Thigh circumference at Week 12 | Week 12 (Evaluated weekly at physical therapy visits from 0-12 weeks)
  Measurement of thigh circumference (centimeters) will be performed utilizing tape measures at specified distances along the thigh

SECONDARY OUTCOMES:
International Knee Documentation Committee (IKDC) Score at Week 6 | 6 weeks (measured at 6 weeks, 3 months, and 6 months post-operatively)
  Patient-reported outcome measure (numerical score) from survey. Min: 0 = lowest level of function/highest level of symptoms. Max: 100 = highest level of function/lowest level of symptoms
International Knee Documentation Committee (IKDC) Score at Week 12 | 3 months (measured at 6 weeks, 3 months, and 6 months post-operatively)
  Patient-reported outcome measure (numerical score) from survey. Min: 0 = lowest level of function/highest level of symptoms. Max: 100 = highest level of function/lowest level of symptoms
International Knee Documentation Committee (IKDC) Score at Week 24 | 6 months (measured at 6 weeks, 3 months, and 6 months post-operatively)
  Patient-reported outcome measure (numerical score) from survey. Min: 0 = lowest level of function/highest level of symptoms. Max: 100 = highest level of function/lowest level of symptoms
Y-balance testing at Week 12 | 3 months (performed at 3 months and 6 months post-operatively)
  Functional outcome measure (numerical score). The lower quarter Y-balance test evaluates dynamic stability and functional symmetry. The subject stands on a single leg and reaches in three directions (anterior, posteromedial, posterolateral) and a composite score is calculated as a percentage: (sum of reach distances in each direction) / (3*limb length) * 100.
Y-balance testing at Week 24 | 6 months (performed at 3 months and 6 months post-operatively)
  Functional outcome measure (numerical score). The lower quarter Y-balance test evaluates dynamic stability and functional symmetry. The subject stands on a single leg and reaches in three directions (anterior, posteromedial, posterolateral) and a composite score is calculated as a percentage: (sum of reach distances in each direction) / (3*limb length) * 100.
3-hop test at Week 12 | 3 months (performed at 3 months and 6 months post-operatively)
  Functional outcome measure (numerical score). The 3-hop test assesses dynamic stability and limb control. The subject hops three times consecutively forward in a same line and at the final landing, pauses in position while a measurement is made from the starting line to the toe at the end of the final hop in centimeters. The test is compared to the contralateral, uninjured limb, and scoring is reported as a percentage of the uninjured limb.
3-hop test at Week 24 | 6 months (performed at 3 months and 6 months post-operatively)
  Functional outcome measure (numerical score). The 3-hop test assesses dynamic stability and limb control. The subject hops three times consecutively forward in a same line and at the final landing, pauses in position while a measurement is made from the starting line to the toe at the end of the final hop in centimeters. The test is compared to the contralateral, uninjured limb, and scoring is reported as a percentage of the uninjured limb.
Single leg squat testing at Week 12 | 3 months (performed at 3 months and 6 months post-operatively)
  Functional outcome measure (numerical score). Single leg squat testing evaluates core stability and ability to perform functional movement safely. Subjects will be asked to perform a single leg squat and will be evaluated on 5 criteria, with one point for clinician-rated good performance in each (A) maintenance in balance, depth, speed (B) trunk posture (C) pelvic rotation & tilt (D) Hip adduction or femoral internal rotation (E) knee joint apparent valgus. Min: 0 = poor balance and motor control; Max: 5 = good balance and motor control
Single leg squat testing at Week 24 | 6 months (performed at 3 months and 6 months post-operatively)
  Functional outcome measure (numerical score). Single leg squat testing evaluates core stability and ability to perform functional movement safely. Subjects will be asked to perform a single leg squat and will be evaluated on 5 criteria, with one point for clinician-rated good performance in each (A) maintenance in balance, depth, speed (B) trunk posture (C) pelvic rotation & tilt (D) Hip adduction or femoral internal rotation (E) knee joint apparent valgus. Min: 0 = poor balance and motor control; Max: 5 = good balance and motor control

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Allahabadi, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No